CLINICAL TRIAL: NCT04488978
Title: A Randomized, Double-blind, Multicenter, Factorial Design, Phase II Study to Evaluate the Efficacy and Safety of Irbesartan and Amlodipine Combined or Alone in Patients With Essential Hypertension
Brief Title: Phase 2 Study to Evaluate the Efficacy and Safety of Irbesartan and Amlodipine Combined or Alone in Patients With Essential Hypetension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Handok Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AI-C201
Record Dates: First submitted 2020-07-21; First posted 2020-07-28 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Irbesartan; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Irbesartan low/Amlodipine low (Experimental): Irbesartan low & Amlodipine low, once daily for 8 weeks
  Interventions: Drug: Irbesartan/Amlodipine
- Irbesartan low/Amlodipine high (Experimental): Irbesartan low & Amlodipine high, once daily for 8 weeks
  Interventions: Drug: Irbesartan/Amlodipine
- Irbesartan high/Amlodipine low (Experimental): Irbesartan high & Amlodipine low, once daily for 8 weeks
  Interventions: Drug: Irbesartan/Amlodipine
- Irbesartan high/Amlodipine high (Experimental): Irbesartan high & Amlodipine high, once daily for 8 weeks
  Interventions: Drug: Irbesartan/Amlodipine
- Amlodipine low (Active Comparator): Amlodipine low, once daily for 8 weeks
  Interventions: Drug: Irbesartan/Amlodipine
- Amlodipine high (Active Comparator): Amlodipine high, once daily for 8 weeks
  Interventions: Drug: Irbesartan/Amlodipine
- Irbesartan low (Active Comparator): Irbesartan low, once daily for 8 weeks
  Interventions: Drug: Irbesartan/Amlodipine
- Irbesartan high (Active Comparator): Irbesartan high, once daily for 8 weeks
  Interventions: Drug: Irbesartan/Amlodipine

INTERVENTIONS:
Drug: Irbesartan/Amlodipine — QID

SUMMARY:
A Randomized, Double-blind, Multicenter, Factorial Design, Phase II Study to Evaluate the Efficacy and Safety of Irbesartan and Amlodipine Combined or Alone in Patients With Essential Hypertension

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 19 years or older / 75 years or younger on screening
* Signed informed consent
* Patients with Essential Hypertension
* Other inclusion applied

Exclusion Criteria:

* Orthostatic hypertension with symptom
* Other exclusion applied

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2021-11-09 (Actual)

PRIMARY OUTCOMES:
The change in MSSBP between baseline and Week8. | Baseline and Week8
  The primary efficacy variable was the change in Mean Sitting Systolic Blood Pressure between baseline and Week8.

SECONDARY OUTCOMES:
The change in MSSBP between baseline and Week4. | Baseline and Week4
The change in Mean Sitting Diastolic Blood Pressure between baseline and Week4 / Week8. | Baseline and Week4/8
The proportion of patients having reached MSSBP < 140 mmHg and MSDBP < 90 mmHg at W4 and at W8. | Baseline and Week4/8

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea